CLINICAL TRIAL: NCT03357549
Title: Effectiveness of an Brief Motivational Intervention to Promote Breastfeeding
Brief Title: Project to Promotion of Breastfeeding
Acronym: MOTIVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Cristina Franco Antonio, Nurse specialist in obstetrics and gynecology (Midwife), University of Extremadura
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Moti003
Record Dates: First submitted 2017-10-23; First posted 2017-11-30 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Breast Feeding
Keywords: Breast Feeding; Motivational Interviewing; Self Efficacy
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Motivational Intervention (Experimental): The women of this group will receive a Brief Motivational Intervention during 20 or 30 minutes.
  Interventions: Other: Brief Motivational Intervention
- Breastfeeding education (Active Comparator): The women of this group will receive a standard education about breastfeeding during 20-30 minutes
  Interventions: Other: Breastfeeding education

INTERVENTIONS:
Other: Brief Motivational Intervention — The Brief Motivational Intervention is an intervention that use strategies are typical of patient-centered interventions. These strategies will help the interviewer to listen, to elicit important information, and to build rapport with the patient and should be used throughout the intervention. The four strategies are Open-Ended Questions, Affirmations, Reflections and Summaries. The objective of de BMI is to increase the client motivation to adopt healthy initiatives, and to increase their self-efficacy to reach their own objectives.
  Arms: Brief Motivational Intervention
Other: Breastfeeding education — It's a common educational intervention about breastfeeding. The women will receive the information by a leaflet with information about breastfeeding and community resources and they will receive verbal information during 20-30 minutes to resolve their doubts.
  Arms: Breastfeeding education

SUMMARY:
Breastfeeding is the ideal feeding for the newborn. The success of the initiation and maintenance of breastfeeding can be influenced by different factors, as breastfeeding self-efficacy. Brief Motivational Intervention (BMI) is a form of collaborative guidance, person-centered approach aimed at strengthening the motivation to adopting healthy initiatives and can increase the self-efficacy.

The hypothesis is that an BMI to promote breastfeeding, during immediate postpartum plus telephone support at the first and third postpartum months, will significant increase in the adherence and duration of breastfeeding compared with the habitual education action applied at the same time. Also, the BMI will increase the breastfeeding self-efficacy of the particpants, and this breastfeeding self-efficacy will be a mediator of the effect between the IMB and the breastfeeding duration.

The general self-efficacy of the participants will change the size of the effect of BMI.

ELIGIBILITY:
Inclusion Criteria:

* All women with term gestations who have given birth healthy newborns by vaginal delivery at the hospital .who agree to participate in the study by signing informed consent, will be includes in the study

Exclusion Criteria:

* Mothers who, by medical indication or own decision, do not initiate breastfeeding in the first hour of the newborn's life.
* Mother of children who require admission to the neonatal unit.
* Women with a previously diagnosed psychiatric disorder.
* Neurological or cognitive impairment that impedes the evaluation and the BMI
* Resident status that prevents correct follow-up of patients (eg. residence outside Spain).
* Women with language or communication barriers

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Changes in degree of exclusivility of Breastfeeding | 1st, 3st and 6th month postpartum
  Breastfeeding is measure acording to degree of exclusivity, acording to WHO definition: Exclusive breastfeeding, Predominant breastfeeding and Partial breastfeeding

SECONDARY OUTCOMES:
Changes in Breastfeeding Self-efficacy | Pre-intervention. 1st, 3rd and 6th month
  Measure with Breastfeeding Self-efficacy Scale-Short Form (BSES-SF). This scale has a maximum score of 70 and a minimum of 14. Higher scores are related to greater maternal self-efficacy in breastfeeding. Breast-feeding self-efficacy is a mother's confidence in her ability to breastfeed and is predictive of breastfeeding behaviors
Changes on General Self-efficacy | Pre-intervention, 1st, 3rd and 6th month
  Measure with General Self-efficacy Scale. This 10-item questionnaire assesses the belief of people about their ability to properly handle stressors of the daily life. This scale has a maximum score of 100 and a minimum of 10. Higher scores are related to greater general self-efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Franco, Midwife, Principal Investigator — Extremadura University
Locations (1):
- Don Benito- Villanueva's Hospital, Don Benito, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Franco-Antonio C, Calderon-Garcia JF, Santano-Mogena E, Rico-Martin S, Cordovilla-Guardia S. Effectiveness of a brief motivational intervention to increase the breastfeeding duration in the first 6 months postpartum: Randomized controlled trial. J Adv Nurs. 2020 Mar;76(3):888-902. doi: 10.1111/jan.14274. Epub 2019 Dec 18. PMID 31782535